CLINICAL TRIAL: NCT05397379
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Safety, Tolerability, Efficacy, and Pharmacokinetics of Orally Administered HEC96719 Tablets in Adult Patients With Presumed Non-Cirrhotic Non-Alcoholic Steatohepatitis
Brief Title: A Safety, Tolerability, Efficacy, and Pharmacokinetics Study of HEC96719 in Subjects With Non-Cirrhotic Non-Alcoholic Steatohepatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC96719-NASH-201
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2022-05

CONDITIONS: Non-Alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- HEC96719 0.25 mg (Experimental): Oral dose once daily for 12 weeks
  Interventions: Drug: HEC96719
- HEC96719 0.35 mg (Experimental): Oral dose once daily for 12 weeks
  Interventions: Drug: HEC96719
- HEC96719 0.5 mg (Experimental): Oral dose once daily for 12 weeks
  Interventions: Drug: HEC96719
- HEC96719 0.25 mg bid (Experimental): Oral dose twice daily for 12 weeks
  Interventions: Drug: HEC96719
- Placebo (Placebo Comparator): Oral dose once or twice daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HEC96719 — Oral tablets
  Arms: HEC96719 0.25 mg; HEC96719 0.25 mg bid; HEC96719 0.35 mg; HEC96719 0.5 mg
Drug: Placebo — Comparator
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled study designed to evaluate the safety, tolerability, efficacy, and pharmacokinetics of HEC96719 in non-cirrhotic NASH patients.

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document must be signed and dated by the subject
* Male or female, 18 to 65 years of age
* Body mass index (BMI)≥18.0 and≤35.0 kg/m2, and Weight≥40 kg;
* Presumed NASH based on clinical characteristics or prior liver biopsy
* MRI PDFF liver fat content ≥ 10 %

Exclusion Criteria:

* previous diagnosis of other forms of chronic liver disease
* Laboratory Screening Results:

  * AST > 5 x ULN
  * ALP > 3 x ULN
  * Total bilirubin > 1.5 x ULN
  * Albumin < 3.2 g/dL
  * INR > 1.3
  * Platelet count < 100,000 /mm3
  * creatinine clearance <60 ml/min (based on Cockroft Gault method)
* previous exposure to OCA
* uncontrolled diabetes mellitus
* presence of cirrhosis
* patients with contraindications to MRI imaging

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | 12 weeks

SECONDARY OUTCOMES:
Mean Change From Baseline in Percentage of Fat in the Liver as Assessed by Magnetic Resonance Imaging - Proton Density Fat Fraction (MRI-PDFF) at Week 12 | Baseline and Week 12
Plasma concentration of HEC96719 - AUC | 4 weeks
  Area under the curve
Plasma concentration of HEC96719 - Cmax | 4 weeks
  Maximum observed concentration
Plasma concentration of HEC96719 - Tmax | 4 weeks
  Time to reach maximum measured plasma concentration
Plasma concentration of HEC96719 - t1/2 | 4 weeks
  Determination of half-life

CONTACTS AND LOCATIONS:
Overall Officials: Jinlin Hou, Doctor, Study Chair — Nanfang Hospital, Southern Medical University
Locations (9):
- China (9):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - NanFang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Affiliated Hospitol of Guangdong Medical University, Guangzhou, Guangdong
  - Union Hospital, TongJi Medical College, HuaZhong University of Science and Technology, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospitol of Xi'an Jiaotong University, Xi’an, Shanxi
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospitol of Wenzhou Medical University, Wenzhou, Zhejiang